CLINICAL TRIAL: NCT01623791
Title: Random Urine Protein-creatinine Ratio to Predict Magnitude of Proteinuria in Different Severity of Pre-eclamptic Patients
Brief Title: Random Urine Protein-creatinin Ratio to Predict Magnitude of Proteinuria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ümran Küçükgöz Güleç, Asist. Prof. Dr, Cukurova University
Other Study IDs: ÇÜTFKHD
Record Dates: First submitted 2012-06-16; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Pre-eclampsia
Keywords: Pre-eclampsia; Proteinuria; Protein - creatinine ratio; Dipstick proteinuria; Severity of disease
MeSH Terms: conditions — Pre-Eclampsia; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — URINE
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Group 1: mild pre-eclamptic group Mild and severe pre-eclampsia were defined American College of Obstetrics and Gynecology criteria (ACOG practice bulletin no. 33: diagnosis and management of preeclampsia and eclampsia. January 2002.)
- Group 2: Group 2: severe pre-eclamptic group

SUMMARY:
The aim of this study was to evaluate diagnostic accuracy of the spot urinary proteinuria, random urine protein- creatinin ratio for prediction of significant proteinuria (≥ 300 mg/24h) and magnitude of proteinuria in patients with in mild preeclampsia and severe preeclampsia. The cross-sectional longitudinal study design used, 209 patients with pre-diagnosed preeclampsia in which in our inpatients clinic included this study. Random urine samples were taken before the 24 hour urine collection for spot urine analysis for evaluated proteinuria and protein/creatinin ratio. 24 hour urine analysis was performed in all patients as the gold standard of the urine total proteinuria.

DETAILED DESCRIPTION:
Group 1 consisted of mild preeclampsia and gestational preeclamptic patients and group 2 consisted of severe preeclamptic patients. The predictive values of the spot urinary dipstick proteinuria and protein/creatinin ratio were determinant and the correlations of the diagnostic test of 24 hour total proteinuria were evaluated. The correlations of the severity of the disease and the tests of the proteinuria were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 16-50 years old, > 20 gestational week pregnant women pre-diagnosed preeclampsia.
* Diagnosis and follow-up performed in inpatients clinic.

Exclusion Criteria:

* The history of chronic hypertension
* The history of systemic illness such as pre-gestational diabetes, systemic lupus erythematosis , malignancies, renal disease.
* Pre-existing urinary tract infections
* Premature rupture of membranes
* Patients who have previously been enrolled in the study

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients admitted to the University of Cukurova, School of Medicine, Department of Obstetrics and Gynecology between May 2011- May 2012 for evaluation of possible preclampsia and/or characterization of the severity of the preeclampsia were offered participation of this study.
Sampling Method: Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Prediction of significant proteinuria | 24 hour urine collection
  Significant proteiuria:(≥ 300 mg/24h)

SECONDARY OUTCOMES:
Predict to magnitude of total proteinuria | 24 hour
  Total proteinuria/24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Umran Kucukgoz Gulec, Assist.Prof., Principal Investigator — Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Cote AM, Brown MA, Lam E, von Dadelszen P, Firoz T, Liston RM, Magee LA. Diagnostic accuracy of urinary spot protein:creatinine ratio for proteinuria in hypertensive pregnant women: systematic review. BMJ. 2008 May 3;336(7651):1003-6. doi: 10.1136/bmj.39532.543947.BE. Epub 2008 Apr 10. PMID 18403498
- [Derived] Kucukgoz Gulec U, Sucu M, Ozgunen FT, Buyukkurt S, Guzel AB, Paydas S. Spot Urine Protein-to-Creatinine Ratio to Predict the Magnitude of 24-Hour Total Proteinuria in Preeclampsia of Varying Severity. J Obstet Gynaecol Can. 2017 Oct;39(10):854-860. doi: 10.1016/j.jogc.2017.04.035. Epub 2017 Jun 21. PMID 28647444